CLINICAL TRIAL: NCT01377207
Title: Optical Coherence Tomography Assessment of Gender diVersity In Primary Angioplasty. The OCTAVIA Trial
Acronym: OCTAVIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Italian Society of Invasive Cardiology (Other)
Collaborators: Meditrial SrL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27/01/2011
Record Dates: First submitted 2011-01-25; First posted 2011-06-21 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Acute Myocardial Infarction
Keywords: ST segment Elevation Myocardial Infarction; Optical Coherence Tomography; Percutaneous Coronary Intervention; Thrombus hystopathology; Gender differences
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Female Arm (Experimental): Female gender diagnosed with ST segment Elevation Myocardial Infarction (STEMI)
  Interventions: Procedure: Primary PCI
- Male Arm (Active Comparator): Male Gender diagnosed with ST segment Elevation Acute Myocardial Infarction (STEMI)
  Interventions: Procedure: Primary PCI

INTERVENTIONS:
Procedure: Primary PCI — Thrombus aspiration and hystopathological analysis, Optical Coherence Tomography assessment of STEMI culprit vessel, Primary PCI with Drug Eluting Stent implantation; Repeat OCT assessment of culprit vessel at 9 monts follow-up

SUMMARY:
Recent studies suggest important gender differences in the pathophysiology and prognosis of ST-segment elevation myocardial infarction (STEMI). This is the first prospective controlled study to assess gender differences in the mechanism of plaque rupture/erosion and thrombus formation in patients presenting with STEMI treated with primary angioplasty. Gender-related mechanisms of plaque rupture or erosion will be investigated using a combination of Quantitative Coronary Angiography, high resolution Optical Coherence Tomography of the culprit vessel and histopathologic analyses of thrombus aspirates of the infarct related lesion, performed by independent core laboratories, blinded to group (male or female) and clinical variables.

DETAILED DESCRIPTION:
In OCTAVIA; enrollment in a 1:1 ratio according to gender group will be ensured by a computer-assisted matching algorithm for gender and age (< 50, 51-70, and > 70 years). Matching has the purpose to enable enrollment of an even number of male and female patients in balanced age groups. This type of dynamic algorithm is appropriate when the composition of the referral population is not known in advance.

OCTAVIA will assess gender differences in the mechanism of plaque rupture. The study will also evaluate the changes in the vascular territory remote from the infarct related lesion, the local vascular response to primary angioplasty interventions and the correlation with clinical outcomes over one year of follow-up. These data are important to support a gender based differential strategy and can have a substantial impact for the improvement of clinical practice in the treatment of women with STEMI.

The study sample of 140 patients is sized to address the hypothesis that the female population has a lower prevalence of plaque rupture (primary endpoint) at baseline OCT than the male population. Computations were conducted assuming a prevalence of rupture of 82% in males and 60% in female patients (22% lower).

Confirmatory power calculation was performed on the basis of stent Strut Coverage at 9 month follow-up (co primary endpoint). Stent-strut coverage and apposition have been linked to the risk of stent thrombosis. However, our understanding of DES healing in male and female patients with ST-segment elevation myocardial infarction is restricted to post-mortem data. The investigators assumed a per patient stent strut coverage (a continuous variable with right skewed distribution) with mean of 97.0% and standard deviation of 4.0% in men, versus mean of 95.0% and standard deviation of 4.0% in women, following Xience Prime implantation. Thus, aiming for a 5% 2-tailed superiority alpha, an 80% power, and assuming a 1:1 enrollment according to gender, a total of 64 patients per group should be enrolled. Anticipating a 10% dropout rate due to patients lost to follow-up and inadequate imaging (included major side branch sections), the total enrollment is set at 70 patients per group (total population of 140 subjects).

ELIGIBILITY:
Inclusion Criteria:

* Acute Myocardial MI with ST segment Elevation, within 6 hours from symptoms onset
* Native coronary artery disease (no prior stent implant, no prior brachytherapy)
* Signed patient informed consent

Exclusion Criteria:

* Patients with left main disease
* infarct lesions in bypass grafts
* cardiogenic shock
* renal failure
* recent major bleeding
* allergy to aspirin or clopidogrel
* on anticoagulant therapy
* no suitable anatomy for OCT (extreme tortuousity, very distal culprit lesion, and large infarct vessel > 4 mm in diameter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Percentage of ruptured or eroded plaques at infarct related lesion as assessed by OCT before PCI | Plaque rupture is evaluated during the index PCI procedure.
  To assess gender differences in the percentage of ruptured or eroded plaques at infarct related lesion as assessed by OCT. The OCT measurement is taken before stenting, when a TIMI flow 2-3 is detected. If baseline flow is TIMI 1, thrombus aspiration is performed before OCT.
Percent of covered stent struts by OCT in infarct-related lesion at 9 months (co-primary endpoint). | Stent coverage is evaluated at 9 months by OCT performed in all patients.
  To assess gender differences in the percentage of covered stent struts at infarct related lesion as assessed by OCT performed in all patients at 9 months.

SECONDARY OUTCOMES:
Minimal Fibrous Cap Thickness (MFCA) (µm) at infarct-related lesion as determined by OCT. | MFCA at index procedure (immediately after reestablishment of TIMI 2-3 coronary flow by PCI) and at 9 months OCT performed in all patients.
  To assess gender differences in Minimal Fibrous Cap Thickness at infart related lesion by OCT immediataly after reestablishment of TIMI (Thrombolysis In Myocardial Infarction) 2-3 coronary blood flow and before stent implantation.
  The evolution of fibrous cap thickness over time will be determined by OCT that will be performed in all patients at 9 months from the index procedure.
Presence and type of residual thrombus material in the culprit vessel. | Residual thrombus in the infarct related vessel is evaluated during the index procedure: immediately after reestablishment of TIMI 2-3 coronary flow during primary percutaneous coronary intervention
  To assess gender differences in thrombus type by OCT in culprit vessel after reestablishment of TIMI (Thrombolysis In Myocardial Infarction) 2-3 coronary blood flow and before stent implantation.
Number of TCFA (<65 µM) as assessed by OCT in the culprit vessel (infarct related). | Thin Fibrous Cap Atheroma is assessed during the index procedure: immediately after reestablishment of TIMI 2-3 coronary flow before stent implantationduring PCI; and at 9 months by OCT performed in all patients.
  To assess gender difference in TCFA number as assessed by OCT in the infarct related vessel during the index procedure and at 9 months by OCT performed in all patients
percent of malapposed-uncovered struts | 9 months
  to assess gender difference in % malapposed/uncovered struts at 9 months follow up by OCT
percent net volume obstruction | 9 months
  To assess gender difference in % of stent volume obstruction by OCT at 9 months follow up
percent abnormal intraluminal tissue | 9 months
  To assess gender difference in % of abnormal intraluminal tissue by OCT at 9 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Guagliumi, MD, Principal Investigator — Italian Society of Invasive Cardiology
Locations (14):
- Italy (14):
  - Ospedale Cardinal Massai, Asti, AT
  - Ospedali Riuniti di Bergamo, Bergamo, BG
  - Policlinico S.Orsola- Malpighi, Bologna, BO
  - Ospedale Ferrarotto, Catania, CT
  - Ospedale S. Anna, Ferrara, FE
  - USL 9 Grosseto, Grosseto, GR
  - Policlinico Gemelli, Rome, Italy
  - Policlinico Padova, Padua, PD
  - Policlinico Parma, Parma, PR
  - Policlinico Le Scotte, Siena, SI
  - Ospedale San Giovanni Bosco, Torino, TO
  - Ospedale Le Molinette, Torino, TO
  - Ospedale Mauriziano, Torino, TO
  - Ospedale Civile, Mirano, VE

REFERENCES:
- [Derived] Saia F, Komukai K, Capodanno D, Sirbu V, Musumeci G, Boccuzzi G, Tarantini G, Fineschi M, Tumminello G, Bernelli C, Niccoli G, Coccato M, Bordoni B, Bezerra H, Biondi-Zoccai G, Virmani R, Guagliumi G; OCTAVIA Investigators. Eroded Versus Ruptured Plaques at the Culprit Site of STEMI: In Vivo Pathophysiological Features and Response to Primary PCI. JACC Cardiovasc Imaging. 2015 May;8(5):566-575. doi: 10.1016/j.jcmg.2015.01.018. Epub 2015 Apr 15. PMID 25890582
- [Derived] Guagliumi G, Capodanno D, Saia F, Musumeci G, Tarantini G, Garbo R, Tumminello G, Sirbu V, Coccato M, Fineschi M, Trani C, De Benedictis M, Limbruno U, De Luca L, Niccoli G, Bezerra H, Ladich E, Costa M, Biondi Zoccai G, Virmani R; OCTAVIA Trial Investigators. Mechanisms of atherothrombosis and vascular response to primary percutaneous coronary intervention in women versus men with acute myocardial infarction: results of the OCTAVIA study. JACC Cardiovasc Interv. 2014 Sep;7(9):958-68. doi: 10.1016/j.jcin.2014.05.011. Epub 2014 Aug 13. PMID 25129664